CLINICAL TRIAL: NCT01442233
Title: Randomized Clinical Trial of Plasma Exchanges Versus Sham Plasma Exchanges in Disabling Multiple Sclerosis Acute Relapses Refractory to Steroid Treatment
Brief Title: Plasma Exchanges in Multiple Sclerosis (MS) Relapses
Acronym: PLASMASEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2010/46
Record Dates: First submitted 2011-08-09; First posted 2011-09-28 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Acute Relapsing
Keywords: multiple sclerosis; plasma exchange
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Plasma Exchange

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plasma exchange (Experimental): 6 plasma exchanges during 2 weeks after randomization
  Interventions: Procedure: plasma exchange
- sham exchange (Sham Comparator): 6 sham plasma exchanges during 2 weeks after randomization
  Interventions: Procedure: sham exchanges procedure

INTERVENTIONS:
Procedure: plasma exchange — 6 plasma exchange each 48 hours during 2 weeks after randomization
  Arms: plasma exchange
Procedure: sham exchanges procedure — 6 sham exchanges each 48 hours during 2 weeks after randomization
  Arms: sham exchange

SUMMARY:
In more than 40 % of multiple sclerosis (MS) patients experiencing relapse, residual disability accumulates in spite of steroid treatment. Plasma exchanges are frequently used but there is no established evidence of their efficacy.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) relapses are usually treated by steroids but some patients did not respond well to this treatment. In more than 40 % of MS patients experiencing relapses, residual disability accumulates in spite of steroid treatment and did not recover. Plasma exchanges (PE) are frequently used to treat the severe attacks of inflammatory demyelination in the central nervous system resistant to steroids (Tumani, 2008). This strategy has been evaluated so far only in few studies. Only one randomized controlled study has been performed (Weinshenker et al, 1999) including patients with very severe attacks of inflammatory demyelinating diseases of various origin (MS, acute transverse myelitis, acute disseminated encephalomyelitis, neuromyelitis optica), not improved after a treatment by steroids. A moderate or important improvement of incapacity was observed in 8 cases out of 19 (42.1%) after treatment by PE against 1 out of 17 (5.9%) after sham treatment. This study concerned only 12 patients having a relapse of MS. Based on this first controlled study and the experience of treatment of 42 MS patients in the department of Neurology of the University Hospital Pellegrin (CHU de Bordeaux) we designed a randomized controlled study of PE against sham PE in moderate to severe acute exacerbations of MS not responding to steroid treatment.

The purpose is to compare plasma exchanges versus sham exchanges on residual disability in MS patients with a demyelinating inflammatory episode (MS or syndrome with high risk of MS) experiencing a disabling relapse not improved after steroid treatment. The primary end-point will be evaluated one month after start of therapy. Secondary endpoints include safety and evaluation of improvement at 3 and 6 months and evaluation of safety

ELIGIBILITY:
Inclusion Criteria:

* Probable relapsing-remitting MS (RRMS) according to Polman et al criteria 2010. or clinically isolated neurological syndrome (CIS) compatible with a demyelinating inflammatory episode within the central nervous system, potentially beginning multiple sclerosis (MS).
* Age 18-65
* EDSS before the current relapse <6.5
* Acute relapse (optic neuritis, motor pyramidal relapse, cerebellar relapse, oculomotor relapse) since less than 2 months
* Having been treated by IV or orally steroid (Methylprednisolone, 1g/d for at least 3 days), followed or not by oral tapering.
* The current relapse inducing a significant clinical deterioration as compared to pre-relapse status and persisting 30 days after starting steroids.

  * Loss of visual acuity more than 30% on one ot both eyes;
  * Or: increase of 1 point pyramidal or brainstem functional system score (FSS) (if score ≥ 3) or cerebellar FSS (if score ≥ 2).
  * Or: reduced walking distance associated with an increase ≥ 0.5 point EDSS if EDSS ≥4.0;
* Having signed informed consent.
* affiliated to the French Social Security

Exclusion Criteria:

* Infection
* Improving relapse.
* Other disease interfering with evaluation.
* Current treatment by immunosuppressive drug (as cyclophosphamide and mitoxantrone) or interrupted for less than 3 months.
* Modification of DMT since less than 1 month.
* Physical or psychic disease interfering with evaluation or consent.
* Participation to another trial in the last 3 months.
* Inability to establish peripheral central intravenous access;
* Cerebral, autonomic, cardiac or other conditions with increased risk from hypovolemia
* Pregnancy or breast-feeding.
* Woman in age to procreate without effective contraception
* Treatment by monoclonal antibody.
* Progressive course of MS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
4 graded-scale of improvement based on objective scales and functional assessment after 1 month | after 1 month

SECONDARY OUTCOMES:
4 graded-scale of improvement based on objective scales and functional assessment | after 3 months and 6 months
change in functional evaluation by visual analogic scales (VAS) | after 1 month, 3 and 6 months
change in functional scores (kurtzke FS) | after 1 month, 3 and 6 months
change of EDSS scores | after 1 month, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda WITTKOP, MD PhD, Study Chair — university bordeaux hospital; Bruno BROCHET, MD, Study Director — University Hospital Bordeaux, France; Bruno BROCHET, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (6):
- France (6):
  - Service de Neurologie - Hôpital Pellegrin - CHU de Bordeaux, Bordeaux
  - Service de neurologie - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Service de Neurologie - CHRU de Lille, Lille
  - Service de Neurologie - CHU de nancy, Nancy
  - Service de neurologie - CHU de Nantes, Nantes
  - Service de Neurologie - CHU de Starsbourg, Strasbourg